CLINICAL TRIAL: NCT00793169
Title: Serum Concentration of Lidocaine After Local Injection During Mohs Micrographic Surgery
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Other Study IDs: MA-stu1404
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: squamous cell carcinoma of the head or neck
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lidocane: Patients undergoing Mohs micrographic surgery of the face or neck will have their blood drawn before, during, and after the procedure.
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Serum levels were measured

SUMMARY:
The primary objective of this study is to (1) determine whether local injection of lidocaine used during Mohs surgery will elevate serum lidocaine concentrations to a level that could cause systemic symptoms and (2) determine whether sustained high levels of serum lidocaine occur after intralesional anesthesia on the face and neck. This study is a cross-sectional study of 10 subjects with basal cell carcinoma or squamous cell carcinoma of the face or neck requiring Mohs micrographic surgery. The study will consist of a brief questionnaire and blood draws during their Moh's surgical procedure.

ELIGIBILITY:
Inclusion Criteria

* Age: 18-75
* Basal cell carcinoma or squamous cell carcinoma of the head or neck
* Subjects are in good health
* Subjects that have the willingness and the ability to understand and provide informed consent for the use of their blood and communicate with the investigator

Exclusion Criteria

* Lidocaine sensitivity
* Bleeding disorder
* Pregnancy
* Medical conditions which would impair hepatic blood flow: congestive heart failure, liver dysfunction, peripheral vascular disease.
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a cross-sectional study of 20 subjects with basal cell carcinoma or squamous cell carcinoma of the face or neck requiring Mohs micrographic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Alam M, Ricci D, Havey J, Rademaker A, Witherspoon J, West DP. Safety of peak serum lidocaine concentration after Mohs micrographic surgery: a prospective cohort study. J Am Acad Dermatol. 2010 Jul;63(1):87-92. doi: 10.1016/j.jaad.2009.08.046. Epub 2010 May 11. PMID 20462662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged 18 years and older presenting to the university for Mohs micrographic surgery for removal of basal cell or cutaneous squamous cell carcinoma of the head and neck were eligible for enrollment.
Groups:
- Detectable Lidocaine Concentrations at Each Blood Draw: The number of subjects with detectable serum lidocaine concentrations (<0.1 ug/mL) at each blood draw.
Period: Overall Study
Arm/Group | Detectable Lidocaine Concentrations at Each Blood Draw
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Detectable Lidocaine Concentrations at Each Blood Draw
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 60 [42 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Detectable Serum Lidocaine Concentrations (<0.1 ug/mL) at Each Blood Draw.
Time Frame: 6 hours
Population: Analysis was per protocol.
Measure: Number; unit: Participants
Arm/Group | Detectable Lidocaine Concentrations at Each Blood Draw
Number analyzed (Participants) | 19
Participants
  Blood Draw 1 | 0
  Blood Draw 2 | 1
  Blood Draw 3 | 0
  Blood Draw 4 | 2
  Blood Draw 5 | 1
  Blood Draw 6 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Detectable Lidocaine Concentrations at Each Blood Draw
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Detectable Lidocaine Concentrations at Each Blood Draw (N=19)
Headache (Surgical and medical procedures) | 1 (1) — A patient reported a headache after the first Mohs micrographic surgery stage.
Shaky (Surgical and medical procedures) | 1 (1) — A patient reported feeling shaky after the first Mohs micrographic surgery stage.

LIMITATIONS AND CAVEATS:
Serum rather than plasma lidocaine levels were measured. For lidocaine levels, plasma and serum levels are similar, and serum levels are more routinely reported by reference laboratories. Hence our selection of serum levels for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No